CLINICAL TRIAL: NCT00964366
Title: Two-week Study to Determine and Compare the Tolerance and Irritation Potential of Clindamycin and Benzoyl Peroxide to Dapsone Gel Topical Acne Medications
Brief Title: Study to Determine and Compare the Tolerance and Irritation Potential of Topical Acne Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114545; C0000-408
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; Dapsone; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clindamycin/BPO gel (Experimental): Once-daily applications of clindamycin/BPO gel to the randomized side of the face either left or right.
  Interventions: Drug: clindamycin and benzoyl peroxide
- Dapsone gel (Active Comparator): Twice-daily applications of dapsone gel to one side of the face.
  Interventions: Drug: Dapsone gel

INTERVENTIONS:
Drug: clindamycin and benzoyl peroxide — Daily applications, to the randomized side of the face either left or right, of clindamycin and benzoyl peroxide
  Other Names: Duac® gel
  Arms: Clindamycin/BPO gel
Drug: Dapsone gel — Twice-daily applications of dapsone gel
  Other Names: ACZONE® (dapsone) Gel; 5%
  Arms: Dapsone gel

SUMMARY:
This is a randomized, half-face study. On 1 side of the face, the subject will apply 1 of the 2 test products, clindamycin and benzoyl peroxide or dapsone gel and the contra lateral side of the face will remain non-treated to serve as a control.

DETAILED DESCRIPTION:
This is a single-blind (blinded expert grader), parallel group, randomized, half-face study being conducted at one clinical site. On 1 side of the face, the subject will apply 1 of the 2 test products, clindamycin and benzoyl peroxide or dapsone gel and the contra lateral side of the face will remain non-treated to serve as a control. Approximately 25-30 male and female healthy subjects without facial acne, aged 18 to 45, will be randomly assigned to each product.

The eligible subjects who qualify will be entered into a 2-week treatment phase. The first of application of the study medication will be supervised at the site, Monday through Friday of each week. Any additional applications should be applied by the subjects at home each evening and the times of application recorded on a diary card. Subjects will apply the study product at home on Saturdays and Sundays and record the times of application on a diary card.

A blinded expert grader will rate comparative product tolerance during the study before study product is applied.

Instrumentation measurements of TEWL will be utilized to evaluate product mildness.

Duplicate sebum samples will be taken from the left and right forehead areas and assessed.

Subject will complete questionnaires and all adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
* Male and female subjects aged from 18 to 45 years at time of consent.
* Has a Fitzpatrick Skin Type of I, II, or III.
* Is willing to discontinue use of all facial products (other than the cleanser provided and makeup or razor and facial shave product) on the face for the 3 days before their baseline/day 0 visit and use only the provided facial products and their normal makeup or razor and facial shaving product for the duration of the study.
* Is willing to not change brands of makeup or razor and facial shave product during the study.
* Is willing to refrain from using any facial product on the face other than study products and their normal makeup or razor and facial shave product for the duration of the study.
* Is willing to refrain from exercising prior to their instrument appointments.
* Is willing to refrain from showering or drinking caffeinated beverages within 1 hour prior to their instrument visits.
* Is willing to report to the site for each visit with a clean face and no makeup.
* Is willing to avoid sunburn, tanning, tanning beds or other excessive sun exposure. Understands that if their skin tone changes significantly during the study it will be necessary to discontinue their participation.
* Able to complete the study and to comply with study instructions.
* Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses.

Exclusion Criteria:

* Female subjects who are pregnant, trying to become pregnant, or breast feeding.
* Male subjects that have facial beards (mustache and/or goatee is acceptable).
* Is a Type I diabetic.
* Has active or chronic skin allergies.
* Has a history of acute or chronic disease that might interfere with, or increase the risk of study participation.
* Has participated in other facial studies in the preceding 30 days or other clinical studies in preceding 14 days.
* Had skin cancer treatment in preceding 12 months.
* Has damaged skin on facial areas (eg, from sunburn, tattoos, scars).
* Had any medical procedure (e.g., laser resurfacing, chemical peels, plastic surgery) to facial areas in preceding 12 months.
* Had any cosmetic procedure (e.g., microdermabrasion, etc.) to facial areas within 8 weeks of the baseline visit.
* Use of topical retinoids or related agents for the treatment of acne or photoaging in the preceding 6 months.
* Live in the same household as currently enrolled subjects.
* Employees of investigator/clinical research organization (CRO) or Stiefel Laboratories involved in the study, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.
* Any other condition or factor the investigator or his duly assigned representative believes may affect the skin response or the interpretation of the test results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- cyberDERM, Broomall, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research center. Subject recruitment occurred from July 16, 2009 to Aug. 11, 2009
Pre-assignment Details: Panelists who met the eligibility criteria and were willing to participate in the study were required to undergo a 3-day pre-trial conditioning period where they had to stop the use of all facial products. Panelists were required to use the provided Soap Free Cleanser (SFC) for washing their face and were allowed to apply their normal makeup.
Groups:
- Clindamycin and BPO Gel: Daily applications of Clindamycin and benzoyl peroxide gel to one-half of the face. Clindamycin and benzoyl peroxide facial gel was applied daily to one side of the face of all subjects in this group in a split-face model. On weekdays during the two-week trial, the investigator scored Erythema on a scale of 0 (none) to 8 (severe) and Dryness on a scale of 0 (none) to 8 (severe).
- Dapsone Gel: Twice-daily applications of dapsone gel to one-half of the face. Dapsone facial gel was applied twice daily to one side of the face of all subjects in this group in a split-face model. On weekdays during the two-week trial, the investigator scored Erythema on a scale of 0 (none) to 8 (severe) and Dryness on a scale of 0 (none) to 8 (severe).
Period: Overall Study
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Started | 28 (27 of the 28 enrolled were eligible after screening.) | 25
Completed | 27 | 24
Not Completed | 1 | 1
Not completed — Did not qualify at Day 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Skin Erythema (Redness)
Description: Assessment of erythema as part of an evaluation of tolerance of two treatments: clindamycin and benzoyl peroxide or dapsone gel. This was done by visual assessment by an independent blinded grader using the grading scale shown below.
  Grade Description 0 None 2 Mild erythema 4 Moderate confluent erythema 6 Marked erythema with some edema 8 Marked erythema, edema, possible erosion
Time Frame: 2 Weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Number analyzed (Participants) | 27 | 25
Units on a scale
  Baseline | 1.06 (0.79) | 1.18 (0.63)
  Day 1 | 1.26 (.76) | 1.34 (.81)
  Day 2 | 1.55 (.84) | 1.33 (.85)
  Day 3 | 1.32 (.63) | 1.50 (.59)
  Day 6 | 1.30 (.75) | 1.65 (.92)
  Day 7 | 1.64 (1.02) | 1.53 (.82)
  Day 8 | 1.80 (.80) | 1.60 (.93)
  Day 9 | 1.67 (.95) | 1.45 (.89)
  Day 10 | 1.81 (.89) | 1.85 (1.13)
  Day 13 | 1.52 (1.20) | 1.65 (1.05)
  Day 14 | 2.10 (1.09) | 1.90 (1.15)
Statistical Analysis 1: Comparison: Clindamycin and BPO Gel vs Dapsone Gel; Test type: Superiority or Other; p > 0.05, Dunn's Multiple Comparisons Test

2. Secondary Outcome: Transepidermal Water Loss (TEWL)
Description: To assess skin moisture and hydration using transepidermal water loss (TEWL). These tables record the data obtained for each panelist at Baseline, and on Days 3, 7 and 14 or upon early termination of site(s), if applicable. Results are measured on a continuous scale.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: TEWL rates (gm/m2/hr)
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Number analyzed (Participants) | 27 | 25
TEWL rates (gm/m2/hr)
  Baseline | 10.29 (3.06) | 10.4 (2.93)
  Day 3 | 12.34 (4.80) | 11.21 (3.26)
  Day 7 | 14.39 (3.73) | 11.53 (3.09)
  Day 14 | 13.88 (3.70) | 11.26 (3.08)

3. Primary Outcome: Skin Dryness
Description: The amount of dryness on the left and right cheek of each panelist.
  The scale used to evaluate skin dryness is:
  Grade Description 0 None 2 Slight flaking 4 Moderate flaking/scaling 6 Marked scaling / slight fissuring 8 Severe scaling, fissuring
  Expert Grader assessments of dryness were taken prior to product application on Days 0, 1, 2, 3, 6, 7, 8, 9, 10, 13 and 14.
Time Frame: Baseline, Day 1through Day 14
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Number analyzed (Participants) | 27 | 25
Units on a scale
  Baseline | 0.11 (0.32) | 0.12 (0.33)
  Day 1 | 0.04 (0.05) | 0.28 (0.71)
  Day 2 | 0.10 (0.26) | 0.23 (0.57)
  Day 3 | 0.16 (0.32) | 0.48 (0.81)
  Day 6 | 0.27 (0.79) | 0.37 (0.64)
  Day 7 | 0.21 (0.45) | 0.23 (0.47)
  Day 8 | 0.54 (1.03) | 0.17 (0.35)
  Day 9 | 0.5 (1.04) | 0.10 (0.20)
  Day 10 | 0.57 (0.91) | 0.15 (0.44)
  Day 13 | 0.57 (1.24) | 0.17 (0.45)
  Day 14 | 0.55 (1.11) | 0.12 (0.28)
Statistical Analysis 1: Comparison: Clindamycin and BPO Gel vs Dapsone Gel; Test type: Superiority or Other; p < 0.05, Dunn's Multiple Comparisons Test — Dapsone versus Clindamycin/BPO gel

4. Secondary Outcome: Sebum Measurements
Description: To sample the skin surface, the sebum collector strips are applied to the skin sites for 10 seconds. Once removed, these samples will be immediately measured for the amount of sebum on the strip using the tape analyzer. The amount of sebum production was measured as the amount of sebum collected on a tape applied to the skin for 10 seconds and then converted to 1 of 10 incremental levels. Sebum production was measured in increments of 0 (minimum value) to 10 (maximum value). The higher the number, the greater amount of sebum produced.
Time Frame: 2 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Number analyzed (Participants) | 27 | 25
units on a scale
  Baseline | 1.72 (1.31) | 2.18 (1.73)
  Day 3 | 1.52 (1.01) | 1.72 (1.11)
  Day 7 | 2.65 (2.05) | 3.33 (2.43)
  Day 14 | 2.35 (2.01) | 2.38 (1.67)
Statistical Analysis 1: Comparison: Clindamycin and BPO Gel vs Dapsone Gel; Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: Skin Hydration
Description: Evaluation of Skin Hydration using electrical conductance measurements,on weekdays during 14 days of treatment. The value recorded which is expressed in units of microsiemens represents the AC conductance 2-3 seconds after placing the spring-loaded probe tip to the sample site.
Time Frame: 2 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Microsiemens
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Number analyzed (Participants) | 27 | 25
Microsiemens
  Baseline | 499.51 (124.27) | 448.31 (149.26)
  4 hours post 1st treatment | 430.38 (156.71) | 404.68 (170.45)
  Day 3 | 614.73 (144.64) | 511.63 (163.97)
  Day 7 | 460.65 (169.03) | 456.73 (173.07)
  Day 14 | 477.80 (173.40) | 471.13 (194.77)
Statistical Analysis 1: Comparison: Clindamycin and BPO Gel vs Dapsone Gel; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 14 days.
Description: Any study product-related AEs ongoing at the end of the treatment period were followed until they resolve, the condition stabilizes, the events are otherwise explained, or the subject is lost to follow-up. In addition, all SAEs were followed until resolution as previously stated for study product-related AEs.
Arm/Group | Clindamycin and BPO Gel | Dapsone Gel
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 2/27 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin and BPO Gel (N=27) | Dapsone Gel (N=25)
Headache (Nervous system disorders) | 1 (1) | 1 (1) — One subject on the clinicamycin/BPO arm was reported to have a headache and one subject on the dapsone arm was reported to have a migrane headache. Neither of these was reported as being related to the study drug by the investigator.
Infection (Infections and infestations) | 1 (1) | 1 (1) — One subject had a urinary tract infeaction in the dapsone treatment group and one subject had a vaginal yeast infection on the clindamycin/ BPO treatment group. Neither of these was reported as being related to the study drug by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days